CLINICAL TRIAL: NCT06761261
Title: Acute Hepatitis in Pediatrics
Acronym: LIVERPED
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: LIVERPED
Record Dates: First submitted 2024-12-01; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-09

CONDITIONS: Hepatitis
Keywords: Hepatitis
MeSH Terms: conditions — Hepatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate wich symptoms and blood test characteristics acute hepatitis manifests in pediatric age. The study will be conducted because acute hepatitis is not an easily and clearly recognized disease in children.

This study aims to better characterize this disease by describing the frequency of the different symptoms with which it can manifest and the changes it causes in blood tests. It also aims to assess the occurrence of any complications of pediatric acute hepatitis.

The study is observational, so it is limited to collecting data and analyzing the patient's clinical course without interfering with normal clinical practice.

DETAILED DESCRIPTION:
Acute hepatitis can be caused by a wide variety of agents, infectious and noninfectious, and vary in severity, from asymptomatic and self-limiting pictures to aggressive and fulminant forms associated with acute liver failure (ALF) that may require liver transplantation. Sometimes acute hepatitis is a prelude to mechanisms of chronic inflammation, with progressive fibrosis, evolution into cirrhosis and liver failure. In cases of hepatocyte damage, the most common laboratory finding is increased transaminases, namely aspartate amino transferase (AST, less specific being present in different tissues) and alanine amino transferase (ALT, more hepatocyte specific). In addition to transaminases, the value of alkaline phosphatase (ALP) and gamma glutamyl transferase (GGT) are useful to better characterize liver damage. An isolated transaminase elevation in an asymptomatic subject is a frequent incidental finding and usually without pathological significance, especially if the increase is less than 2 times the upper limit of normal. Some guidelines (American College of Gastroenterology) recommend confirming the transaminase alteration with a second blood draw and assessing the degree of alteration3; others (British Society of Gastroenterology) recommend targeted investigations regardless of the level of transaminase alteration and duration of hypertransaminasemia: in this case, it is considered more important to carefully consider the clinical context and make a comprehensive assessment of liver function.Acute hepatitis is not always symptomatic, and if it does become symptomatic, the most common signs and symptoms are nonspecific (nausea and vomiting, general malaise, asthenia, anorexia, abdominal pain, jaundice, palpable liver) and do not correlate clearly with the extent of liver parenchyma damage. However, in the presence of acute liver damage, early recognition of progression to ALF is critical because of the associated high mortality, and in such cases refer the patient to a transplant center. ALF is defined as acute liver damage with altered coagulation, expressed as prolongation of the prothrombin time and increased INR, with or without the appearance of signs and symptoms of encephalopathy. In pediatric age, the most frequent causes of ALF are metabolic diseases (in particular, Wilson's disease), viral hepatitis, toxic forms (especially from drugs), and autoimmune forms. There is a lack of recent pediatric studies in the literature investigating the mode of presentation (signs, symptoms, and laboratory changes) of acute liver injury, and highlighting how this presentation varies by age group, depending on the different etiologies at work. Such analysis will be all the more useful considering that acute hepatitis can be clinically subtle and nonspecific, and only by integrating clinic and laboratory tests can it be recognized and diagnostic investigations aimed at recognizing the specific etiology be performed. In addition, the natural history of pediatric acute hepatitis is poorly studied, particularly the possible though rare forms with fulminant course and ALF. The present study aims to describe the clinical presentation and natural history of pediatric acute liver injury from the experience of Pediatric Emergency Room (PSP) units and Pediatrics departments. This would allow a better characterization of an often nonspecific picture, combining clinical and laboratory data, and studying how they change according to age group and different underlying etiologies. In addition, it would allow assessment of the frequency of pediatric ALF in the participating centers.

ELIGIBILITY:
Inclusion Criteria:

* Age between 0 and 17 years (extremes included).
* Access to PSP and/or hospitalized (OBI or hospitalization)
* Diagnosis of acute hepatitis

Exclusion Criteria:

* Refusal of the parent/guardian to participate in the study.
* Mild hypertransaminasemia (<5 times the upper limit of normal) in a patient with known chronic liver dysfunction (e.g. liver cirrhosis).
* Neonatal jaundice without hepatocyte involvement or signs of cholestasis (prevalence of indirect bilirubin with normal AST, ALT and GGT).

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients aged between 0 and 17 years, arriving at the pediatric emergency room and/or admitted to the pediatric ward of the participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 437 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Study the clinical-laboratory presentation of pediatric acute hepatitis and how it varies according to age group and different etiologies. | through study completion, an average of 1 year
  The present study aims to describe the clinical presentation and natural history of pediatric acute liver injury from the experience of Pediatric Emergency Room (PSP) units and Pediatrics departments.
  This would allow a better characterization of an often nonspecific picture, combining clinical and laboratory data, and studying how they change according to age group and different underlying etiologies.
  In addition, it would allow assessment of the frequency of pediatric ALF in the participating centers.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Azienda USL di Bologna Ospedale Maggiore, Bologna
  - IRCCS Azienda Ospedaliero - Universitaria di Bologna, Bologna

IPD SHARING:
Plan to Share IPD: No